CLINICAL TRIAL: NCT00860301
Title: Acupuncture in Infantile Colic - a Randomised Controlled Double Blind Clinical Study
Brief Title: Acupuncture in Infantile Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Ekhagastiftelsen (Other); Magn Bergvalls stiftelse (Unknown); General Maternity Hospital Foundation (Unknown)
Responsible Party: Inger Hallström, Professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-Landgren
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Infantile Colic
Keywords: infantile colic
MeSH Terms: conditions — Colic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture group (Experimental)
  Interventions: Other: Acupuncture
- Control group (No Intervention): Infants come to the clinic six times, are left alone for five minutes with the acupuncture nurse who hold its hand and talks to it.

INTERVENTIONS:
Other: Acupuncture — Infants come to the clinic twice a week for three weeks. Parents meet a nurse and hand the infant to her. The nurse brings the infant to a room where another nurse is alone with the infant for five minutes. Infants in the acupuncture group get acupuncture. One needle is inserted 1-3 mm in the point LI4 on one of the infants hands for one to three seconds and then withdrawn.
  Arms: Acupuncture group

SUMMARY:
The purpose of this study is to investigate whether acupuncture influences:

* the rate of infants who still fulfil the colic criterion after three intervention weeks
* the time when the infants are crying, fussing or have intense bouts of colicky symptoms

DETAILED DESCRIPTION:
Infantile colic is a common problem. Both the baby and the parents are suffering and there is a risk that the early relationship is disturbed. There is no known treatment that is both effective and harmless. Acupuncture releases different neurotransmitters and hormones, gives pain reduction and affects digestion. Acupuncture in infantile colic has not been studied in a scientific way even though the method is used in many countries. In this randomised study we will investigate if acupuncture affects symptoms in infantile colic.

ELIGIBILITY:
Inclusion Criteria:

* 2-8 weeks old otherwise healthy infants who are fussing/crying more than three hours/day, more than three days during one week

Exclusion Criteria:

* infants born before week 36
* infants who dont gain weight properly
* infants taking other medicine than dimethicone or lactobacillus reuteri

Ages: 2 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
If the rate of infants who still fulfil the colic criterion in each of the intervention weeks differ between groups. | First, second and third intervention weeks

SECONDARY OUTCOMES:
If the time when infants are crying, fussing or have intense bouts of colicky symptoms in each of the intervention weeks differ between groups. | First, second and third intervention weeks

CONTACTS AND LOCATIONS:
Overall Officials: Inger Hallström, Professor, Principal Investigator — Lund University
Locations (1):
- Acupuncture Clinic, Helsingborg, Sweden

REFERENCES:
- [Background] Landgren K.& Hallström I. Akupunkturbehandling vid spädbarnskolik - föräldrars upplevelser av barnets beteende före och efter behandling. Vård i Norden, vol.1, 26-31, 2005.
- [Derived] Landgren K, Kvorning N, Hallstrom I. Feeding, stooling and sleeping patterns in infants with colic--a randomized controlled trial of minimal acupuncture. BMC Complement Altern Med. 2011 Oct 11;11:93. doi: 10.1186/1472-6882-11-93. PMID 21989212